CLINICAL TRIAL: NCT03542448
Title: Correlation Between Choroidal Thickness and Myopia Using Swept Source OCT
Brief Title: Choroidal Thickness in Myopes by SSOCT
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Rifaat Mokhtar, Principal investigator, Assiut University
Other Study IDs: ESSO
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: 97 eye of 49 normal Egyptian volunteers were divided into groups according to age, AL, SE of refractive error, minimum corneal thickness (MCT) and mean corneal power as follow:
  Age into 3 groups:
  Group A: from 18 to 30 years old Group B: from 31 to 40 years old Group C: > 40 years old
  Axial length into 3 groups:
  Group A: from 22 to less than 24 mm Group B: from 24 to 26 mm Group C: > 26 mm
  Spherical equivalent of refractive error into :
  Group A : from zero to - 2 D Group B : from - 2 to > - 4 D Group C : from - 4 to > - 6 D Group D: from - 6 to - 8 D
  Minimum corneal thickness (MCT) into 3 groups:
  Group i: < 500 um Group ii: from 500 to 540 um Group iii: > 540 um
  Refractive power of cornea (Mean K) into 3 groups:
  Group 1: 41 to less than 44 D Group 2: 44 to 46 D Group 3: > 46 D
  Interventions: Device: Swept source optical coherence tomography

INTERVENTIONS:
Device: Swept source optical coherence tomography — Measurement of choroidal thickness in myopic patients

SUMMARY:
Optical coherence tomography is a non-invasive and non-contact imaging modality that enables two-dimensional cross-sectional and three-dimensional volumetric imaging of tissue architecture.

DETAILED DESCRIPTION:
It has evolved over the past decade as one of the most important ancillary tests in ophthalmic practice. It is a noninvasive imaging technique and provides high resolution, cross-sectional images of the retina, the retinal nerve fiber layer and the optic nerve head. With axial resolution in the 5-7 μm range, it provides close to an in-vivo 'optical biopsy' of the retina. Optical coherence tomography employs light from a broadband light source, which is divided into a reference and a sample beam, to obtain a reflectivity versus depth profile of the retina. The light waves that are back scattered from the retina, interfere with the reference beam, and this interference pattern is used to measure the light echoes versus the depth profile of the tissue in vivo.

Recently, a new type of optical coherence tomography instrument, called a swept source optical coherence tomography, was introduced. The Swept source optical coherence tomography uses a tunable laser (swept-source) as a light source with a longer wavelength that allows the light to penetrate deeper into tissues than the conventional spectral domain optical coherence tomography instruments. This, then, enabled the imaging of the choroid.

Because choroidal abnormalities such as vascular hyperpermeability, vascular changes, loss and thinning are critical to the onset and progression of many ocular diseases, ophthalmologists and researchers are shifting their interest to the choroidal abnormalities.

Being a major vascular layer of the eye , choroid plays an important role in ocular health, and is involved in the pathogenesis of many intraocular diseases such as age-related macular degeneration , polypoidal choroidal vasculopathy , central serous chorioretinopathy and myopic macular degeneration. Accurate measurement of choroidal thickness in vivo is an essential step in monitoring disease onset and progression that lead to choroidal thinning. Based on histologic study, choroidal thickness ranges from 170 to 220 um.

These disorders show the need for understanding the choroidal structure in ocular diseases and the importance of having database of choroidal thickness.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 years to 40 age.
* Spherical equivalent from zero to -8.
* Minimum corneal thickness from 500 to 540.
* Refractive power of cornea more than 41 diopter.
* Axial length from 22 to 26.

Exclusion Criteria:

* Corneal abnormalities such as ectasia.
* Eyes with dystrophic or degenerative diseases.
* Prior ocular surgery.
* Anterior or posterior segment inflammation.
* Glaucoma.
* Eyes with choroidal abnormalities or conditions that could affect choroidal thickness such as central serous chorioretinopathy, nevus, pregnancy, or haemangiomas.
* Patients with diabetes mellitus.
* Patients with optical media opacity that significantly disturb optical coherence tomography image acquisition.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 100 case of age from 18 to 40 years old of myopic refraction from zero to -8 diopter , minimum corneal thickness from 500 to 540 micrometer , refractive power of cornea more than 41 diopter and axial length from 22 to 26 millimeter
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Comparison between choroidal thickness and myopia | Baseline
  Analysis of choroidal thickness measured by swept source optical coherence tomography and the degree of myopia

CONTACTS AND LOCATIONS:
Locations (1):
- AssiutU, Asyut, Egypt

REFERENCES:
- [Background] Sull AC, Vuong LN, Price LL, Srinivasan VJ, Gorczynska I, Fujimoto JG, Schuman JS, Duker JS. Comparison of spectral/Fourier domain optical coherence tomography instruments for assessment of normal macular thickness. Retina. 2010 Feb;30(2):235-45. doi: 10.1097/IAE.0b013e3181bd2c3b. PMID 19952997